CLINICAL TRIAL: NCT00521040
Title: Evaluation of the Efficacy and Safety of Levocetirizine During 8 Weeks Preceding and Following the Anticipated Onset of the Grass Pollen Season in Subjects Suffering From Seasonal Allergic Rhinitis Associated With Pollen-induced Asthma
Brief Title: Efficacy and Safety of Levocetirizine 8 Weeks Prior and After the Onset of the Grass Pollen Season in Subjects With SAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A00306
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Levocetirizine dihydrochloride; Xyzal tablets
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levocetirizine dihydrochloride

SUMMARY:
Efficacy and Safety of Levocetirizine 8 Weeks Prior and After the Onset of the Grass Pollen Season in Subjects With SAR

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects ≥ 12 years
* 2 year history of seasonal allergic rhinitis
* documented hypersensitivity to local seasonal allergens (grass pollen)
* documented pollen-induced asthma
* without acute ongoing exacerbation of asthma or allergic rhinitis
* no continuous ongoing treatment for rhinitis or asthma

Exclusion Criteria:

* non-allergic rhinitis and anatomic abnormalities disturbing the analysis of nasal capacity
* symptomatic rhinitis or asthma due to tree pollens
* currently treated by specific grass pollen immunotherapy
* suffering from non-allergic asthma
* chronic use of inhaled steroids and/or long acting β2 agonists; and/or corticosteroid dependent asthma
* atopic dermatitis or urticaria requiring an antihistamine treatment or the administration of oral or topical corticosteroids
* contraindication for salbutamol use

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2004-02; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
T4SS (sum of the scores of the severity of sneezing, rhinorrhea, nasal pruritus and ocular pruritus) | 12 weeks

SECONDARY OUTCOMES:
Pollen-induced symptomatology of asthma; symptoms of rhinitis and asthma over the first 4 season weeks and during the entire observation period following the actual onset of the grass pollen season | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma